CLINICAL TRIAL: NCT07398703
Title: "The Impact of Beta-Lactam Infusion Strategy on Treatment Efficacy in Sepsis and Septic Shock : Extended vs. Intermittent Dosing in the ICU"
Brief Title: Extended vs. Intermittent Beta-Lactam Infusion in ICU Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Yousif Sadik Sayed, Resident physician, Assiut University
Other Study IDs: Beta-Lactam Infusion in sepsis
Record Dates: First submitted 2025-09-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sepsis; Septic Shock
Keywords: Beta-lactam; Extended; Intermittent; infusion; Sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Extended infusion of beta-lactam antibiotics
  Interventions: Drug: Extended beta-lactam antibiotics
- Group B: Intermittent infusion of beta-lactam antibiotics
  Interventions: Drug: Intermittent Beta-lactam antibiotics

INTERVENTIONS:
Drug: Extended beta-lactam antibiotics — Group A will be receiving extended infusion of beta-lactam antibiotic over 4 hours.
  Groups: Group A
Drug: Intermittent Beta-lactam antibiotics — Group B will be receiving intermittent infusion of beta-lactam antibiotic over 30 minutes.
  Groups: Group B

SUMMARY:
This observational study compares extended versus intermittent beta-lactam infusion in sepsis patients, assessing survival, clinical cure rates, and practical ICU challenges. The findings will guide optimal antibiotic protocols, potentially improving sepsis outcomes through precision dosing strategies.

DETAILED DESCRIPTION:
Sepsis is defined as a life-threatening organ dysfunction caused by a dysregulated host response to infection. Septic shock should be considered a subset of sepsis in which underlying circulatory, cellular, and metabolic abnormalities significantly increase mortality risk compared to sepsis alone.

Beta-lactam antibiotics exhibit broad-spectrum activity against most Gram-positive and Gram-negative bacteria, making them a key component of sepsis treatment. Their bactericidal effects are time-dependent, meaning efficacy depends on maintaining free drug concentrations above the minimum inhibitory concentration of the target pathogen for an optimal duration.

In clinical practice, beta-lactams are typically administered via intermittent infusion. However, critically ill patients often experience altered pharmacokinetics due to changes in renal clearance, protein binding, fluid balance, and volume distribution. This variability can lead to unpredictable drug concentrations, increasing the risk of subtherapeutic antibiotic exposure.

Existing studies suggest that continuous infusion may enhance beta-lactam efficacy by maintaining drug concentrations above the minimum inhibitory concentration for longer periods, optimizing pharmacokinetic and pharmacodynamic targets. Some meta-analyses and small randomized controlled trials report reduced mortality and improved clinical cure rates with continuous infusion, while others show no significant difference. However, differences in dosing regimens, patient populations, and pharmacokinetic variability in critically ill patients make it difficult to draw firm conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 18 - 65
* Patients admitted to critical care unit diagnosed with pneumonia or urinary tract infection with two of the following:

  1. Temperature: over 38 degree celsius
  2. Heart rate: over 100 beats per minute
  3. Respiratory rate: over 20 breaths per minute
  4. leucocyte count over than 12000 or less than 4000 microlitres or over 10% immature forms or bands
* Patients with positive sputum or urine cultures

Exclusion Criteria:

* Hypersensitivity to Beta-lactams
* Pregnancy
* Very low probability of survival using APAACHE II score > 34 points.
* Immunodeficency or taking immunosuppressive medications
* Acute or chronic renal failure with creatinine clearance less than 30 ml/min according to Cockcroft-Gault formula.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patient diagnosed with pneumonia and urinary tract infection at Critical care unit at Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 90 days from the date of randomization. | Baseline and 90 days

SECONDARY OUTCOMES:
Clinical cure | Baseline and 16 days
  defined as completing the full course of beta-lactam therapy within 14 days without requiring additional antibiotics for the same infection within 48 hours after treatment cessation.

REFERENCES:
- [Background] Dulhunty JM, Roberts JA, Davis JS, Webb SA, Bellomo R, Gomersall C, Shirwadkar C, Eastwood GM, Myburgh J, Paterson DL, Lipman J. Continuous infusion of beta-lactam antibiotics in severe sepsis: a multicenter double-blind, randomized controlled trial. Clin Infect Dis. 2013 Jan;56(2):236-44. doi: 10.1093/cid/cis856. Epub 2012 Oct 16. PMID 23074313
- [Background] Guarino M, Perna B, Cesaro AE, Maritati M, Spampinato MD, Contini C, De Giorgio R. 2023 Update on Sepsis and Septic Shock in Adult Patients: Management in the Emergency Department. J Clin Med. 2023 Apr 28;12(9):3188. doi: 10.3390/jcm12093188. PMID 37176628
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Li X, Long Y, Wu G, Li R, Zhou M, He A, Jiang Z. Prolonged vs intermittent intravenous infusion of beta-lactam antibiotics for patients with sepsis: a systematic review of randomized clinical trials with meta-analysis and trial sequential analysis. Ann Intensive Care. 2023 Dec 5;13(1):121. doi: 10.1186/s13613-023-01222-w. PMID 38051467
- [Background] Tamma PD, Aitken SL, Bonomo RA, Mathers AJ, van Duin D, Clancy CJ. Infectious Diseases Society of America 2023 Guidance on the Treatment of Antimicrobial Resistant Gram-Negative Infections. Clin Infect Dis. 2023 Jul 18:ciad428. doi: 10.1093/cid/ciad428. Online ahead of print. PMID 37463564
- [Background] Povoa P, Coelho L, Dal-Pizzol F, Ferrer R, Huttner A, Conway Morris A, Nobre V, Ramirez P, Rouze A, Salluh J, Singer M, Sweeney DA, Torres A, Waterer G, Kalil AC. How to use biomarkers of infection or sepsis at the bedside: guide to clinicians. Intensive Care Med. 2023 Feb;49(2):142-153. doi: 10.1007/s00134-022-06956-y. Epub 2023 Jan 2. PMID 36592205
- [Background] Mirjalili M, Zand F, Karimzadeh I, Masjedi M, Sabetian G, Mirzaei E, Vazin A. The clinical and paraclinical effectiveness of four-hour infusion vs. half-hour infusion of high-dose ampicillin-sulbactam in treatment of critically ill patients with sepsis or septic shock: An assessor-blinded randomized clinical trial. J Crit Care. 2023 Feb;73:154170. doi: 10.1016/j.jcrc.2022.154170. Epub 2022 Oct 19. PMID 36272277